CLINICAL TRIAL: NCT01969279
Title: Radiographic Influences of Long-term Bisphosphonate Treatment on Femur
Brief Title: Radiographic Influences of Bisphosphonate Treatment on Femur
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tomidahama Hospital (Other)
Responsible Party: Principal Investigator, Toshihiko Kono, Head of Hospital, Tomidahama Hospital
Other Study IDs: IRB TH No 6-2
Record Dates: First submitted 2013-10-13; First posted 2013-10-25 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Femur Fracture
Keywords: Osteoporosis; Bisphosphonate; Atypical femoral fracture; Side effect
MeSH Terms: conditions — Femoral Fractures; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Although there is strong evidence that bisphosphonates prevent certain types of osteoporotic fractures, there are concerns that these medications may be associated with rare atypical femoral fractures (AFF). But the relationship between long-term bisphosphonate treatment and AFF is unclear. In this study, the investigators would like to analyze the long term effects on femur by bisphosphonate treatment.The participants are treated in the investigators hospital more than four years.

DETAILED DESCRIPTION:
Bisphosphonates have been widely used in the treatment of osteoporosis. Recently, long-term use of bisphosphonates increases the risk for AFFs in older women, according to the results of a population-based, nested case-control study. Unique radiographic pattern of AFF is reported, such as simple transverse or short oblique fracture with breaking of medial cortex and cortical thickness. But radiographic evaluation were performed for fracture patients in previous reports and the femoral condition of long-term bisphosphonate treatment patients before fracture is not known.

The main objective of this study is to reveal the effects of long-term bisphosphonate treatment on femur.

ELIGIBILITY:
Inclusion Criteria:

* Patients using bisphosphonate more than four years

Exclusion Criteria:

* patients who could not use bisphosphonate

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oateoporosis patients using bisphosphonate more than four years.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2000-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Influence of long-term bisphosphonate treatment on femur. | Up to 24 month
  The investigators plan to analyze 120 patients who undergo bisphosphonate treatments more than four years.
  We investigate radiographic features in patients with long-term bisphosphonate treatment. We investigate bilateral femur radiographs concerning to cortical thickening and cortical hypertrophy. We also investigate age and sex matched patients without bisphosphonate treatment as a control group.
  To determine the bisphosphonate treatment effects on femur, statistical analyses are performed using Spearman correlation, paired t-test, chi-square test, Fisher's exact test and Mann-Whitney U test. Finally, we conclude the effects of bisphosphonate treatment on femur.

SECONDARY OUTCOMES:
Longitudinal effects of bisphosphonate treatments on femur | Up to108 months
  The investigators plan to analyze 100 patients who undergo bisphosphonate treatments more than four months. To enroll 300 participants including drop-out patients, up to 60 months is required beside 48 months treatment periods.
  In this study, we plan to evaluate longitudinal changes of femur. We evaluate femur radiographs at baseline and every one year. We investigate bilateral femur radiographs concerning to cortical thickening and cortical hypertrophy longitudinally. Statical analyses are performed using Spearman correlation coefficients, paired t-test, Mann-Whitney U test, chi-square test and Fisher's exact test.

CONTACTS AND LOCATIONS:
Locations (1):
- Tomidahama Hospital, Yokkaichi, Mie-ken, Japan